CLINICAL TRIAL: NCT06305988
Title: Neuroregulatory Effect and Mechanism of Transcranial Direct Current Stimulation on Medial Prefrontal Cortex in Autism Spectrum Disorder
Brief Title: Neuroregulatory Effect and Mechanism of tDCS on Medial Prefrontal Cortex in ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jian-Jun Ou (Other)
Responsible Party: Sponsor-Investigator, Jian-Jun Ou, Principal Investigator, Central South University
Organization: Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LYG2023021
Record Dates: First submitted 2024-01-26; First posted 2024-03-12 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: ASD
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group（Transcranial direct current stimulation） (Experimental): tDCS group participants will receive tDCS intervention stimulation for 1 week (1.5mA, 20min/ time, twice a day)
  Interventions: Device: Transcranial direct current stimulation
- control group（Sham Transcranial direct current stimulation） (Placebo Comparator): Placebo comparator group subjects will receive similar sites and the same frequency of spurials (0mA, 20min/ time, twice daily) for 1 week
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — The anode patch is placed in Fz, and the cathode patch is placed on right cheek, powered by direct current with a current of 1.5mA. Subjects in the placebo comparator group will receive sham tDCS for 1 week, which mimics the tDCS intervention in terms of electrode placement and session frequency. However, the device will deliver a 0mA current, ensuring no actual stimulation occurs. The anode patch is placed at Fz, and the cathode patch is positioned on the right cheek, to maintain the blinding of the intervention.

SUMMARY:
In this proposed study, a transcranial direct current stimulator is used to intervene in the medial prefrontal cortex of children with autism, and the efficacy of this intervention method is evaluated, as well as the internal mechanism of Autism Spectrum Disorders' intervention is discussed.

DETAILED DESCRIPTION:
This is a randomized controlled double-blind trial. Using a transcranial direct current stimulator to stimulate the Autism Spectrum Disorders of children with autism, place an anode patch on Fz and a cathode patch on right cheek to observe whether it can improve social and cognitive function in autism. Parameter settings: The current size is 1.5mA. Treat twice a day for 20 minutes, for a total of 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age 4-18 years old;
2. Clinically diagnosed by a psychiatrist with autism spectrum disorder;
3. Confirmed by researchers (pediatric psychiatrists) that they meet the diagnostic criteria for autism spectrum disorders in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) of the United States;
4. Evaluated by researchers (pediatric psychiatrists) using the Autism Diagnostic Interview Revised (ADI-R) and Autism Diagnostic Observation Schedule (ADOS), it is consistent with the diagnosis of autism spectrum disorders;
5. Capable of cooperating with magnetic resonance spectroscopy and transcranial direct current stimulation.

Exclusion Criteria:

* a) Existence of serious physical diseases and conditions, such as significant intracranial lesions, thyroid diseases, epilepsy, congenital heart disease, severe hematological diseases, systemic lupus erythematosus, visual and auditory impairments, etc;

  b) Imaging examination showed significant brain structural abnormalities;

  c) Having serious neurological diseases, a clear family history, or potential risks;

  d) Metal or pacemaker implantation in the body, holes or cracks in the skull;

  e) Taking benzodiazepines or anticonvulsants;

  f) The existence of clear or suspicious genetic diseases;

  g) Conforming to the diagnosis of other serious mental illnesses, such as schizophrenia and bipolar disorder.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Autism assessment assessment index | Baseline, the day after intervention, three weeks after intervention
  3. Autism was assessed using the Oregon State University Autism Rating Scale, DSM-5 (OARS-5), which includes the signs and symptoms of autism spectrum disorders described in the DSM-5. The scores include :1; Total number of symptoms. Every symptom that occurs (i.e., 1, 2, or 3 points) is recorded in the symptom count. 2. Weighted average severity. The clinician scored each item on a scale of 0, 1, 2 or 3 based on the parent's description of the particular problem. 3. Damage index. In Section C of OARS-5, after discussion with the child/adolescent's caregiver, the clinician will rate the level of support on a scale of 0(no support) to 3(maximum support).

SECONDARY OUTCOMES:
EEG physiological detection index | Baseline, the day after intervention, three weeks after intervention
  detect resting state and task state EEG, analyze and calculate the functional E/I ratio of EEG power spectrum
Social Communication Changes index | Baseline, the day after intervention, three weeks after intervention
  Assessed by the Social Response Scale (SRS-II). The change in social communication scores from baseline to the end of the study period will be the primary outcome of interest, the critical value is 59.5, and the total score is the sum of all entries, with the lowest score of 0 and the highest score of 3 for each entry.
Stereotyped behavior index | Baseline, the day after intervention, three weeks after intervention
  The Repetitive Stereotyping Behavior Scale-Revised (RBS-R) is a tool used to assess repetitive and stereotyping behaviors in autism spectrum disorders (ASD) and other related disorders. The scale consists of 5 subscales, namely Ⅰ stereotypical behavior scale, Ⅱ self-injury behavior scale, Ⅲ impulsive behavior scale, Ⅳ ritualistic behavior scale, Ⅴ fixed behavior scale, and the score is 0= these behaviors have never happened -- 3= these behaviors have happened. And it's serious; The number of positive items is items other than those with a zero score.
Sensory index | Baseline, the day after intervention, three weeks after intervention
  The Short Sensory Profile (SSP) was used to assess sensory processing abnormalities in children. Each statement has a rating range, which is a 5-point scale from "always" to "never." Raters need to rate the child based on how often they respond to specific sensory inputs. The total score of the SSP is the sum of the scores of all entries. The lowest score generally reflects a higher level of sensory processing difficulty, while the highest score indicates less difficulty.
Abnormal behavior indicator | Baseline, the day after intervention, three weeks after intervention
  Individuals are assessed for behavioral abnormalities using the Aberrant Behavior Checklist-Second Edition (ABC-II), a scoring system designed according to the frequency and severity of behavioral problems. For each entry, raters are asked to rate it according to the following criteria: 0: no problem at all. Score 1: The behavior is problematic, but the degree is not serious. Score 2: The problem is moderately serious. 3 marks: The problem is serious. The total score for ABC-II is the sum of scores for all entries, with the lowest score (i.e., all entries are rated 0) indicating that no behavioral problems were observed, while the highest score (i.e., all entries are rated 3) indicating widespread and serious behavioral problems.
Sleep index | Baseline, the day after intervention,three weeks after intervention
  Childhood Sleep Disorders Scale (SDSC) was used to assess children's sleep problems and habits. Ratings are usually based on frequency and duration, such as "always," "often," "sometimes," "occasionally," or "never happens." Each entry is typically scored on a scale of 0 to 5, with 0 being no problem and the highest being the most serious. The total score of the CSHQ is the sum of the scores of all entries.

OTHER OUTCOMES:
Plasma Metabolite Levels Assessment | At baseline, the first day of intervention
  The levels of metabolites in plasma will be detected and quantified using a comprehensive Metabolomics detection approach. This method involves analyzing small-molecule chemical compounds found in plasma, providing a broad snapshot of the metabolic state of an organism at the given time points.
Safety evaluation SAFTEE indicator | Baseline, the day after intervention, three weeks after intervention
  The scale is the most commonly used safety assessment tool in clinical trials to assess whether participants had side effects or sudden adverse events during the course of the study. The SAFTEE-GI (General inquiry) version was adopted in this study, which asked subjects in detail whether they had physical or psychological problems, occurrence time, duration, frequency and status quo during a specific period of time, so as to timely discover the adverse reactions of subjects during the clinical trial. Discontinue the study if adverse events occur.

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Ou, doctor, Study Chair — Central South University; Yanting Hou, doctor, Study Director — Central South University
Locations (1):
- Department of Psychiatry, Xiangya Second Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No